CLINICAL TRIAL: NCT00873678
Title: Assessment of the Prevalence and Mutational Spectrum of Genes AHI1, NPHP1 and CEP290 in Joubert Syndrome and Cerebello-oculo-renal Syndromes
Brief Title: Assessment of the Prevalence of Genes AHI1, NPHP1 and CEP290 in Joubert Syndrome
Acronym: JSCORS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel Ouslimani, Department Clinical Research of Developpement
Other Study IDs: P051079
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-03

CONDITIONS: Joubert Syndrome; Cerebello-oculo-renal Syndromes
Keywords: Molar tooth; AHI1 gene; CEP290 gene; ciliopathies
MeSH Terms: conditions — Agenesis of Cerebellar Vermis; Meckel Syndrome, Type 4; Ciliopathies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood sample (10 ml)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children or adult patients affected with JS/CORS
  Interventions: Biological: Whole blood sample

INTERVENTIONS:
Biological: Whole blood sample — Whole blood sample (10 ml)

SUMMARY:
Primary objective:

* assessment of the prevalence of AHI1 mutations in Joubert syndrome and cerebello-oculo-renal syndromes (JS/CORS)

Secondary objective:

* assessment of the prevalence of CEP290 mutations and NPHP1 homozygous deletions in JS/CORS
* caracterization of mutational spectrum of AHI1, NPHP1, CEP290 genes in JS/CORS.
* evaluation of genotype-phenotype correlation in JS/CORS.

DETAILED DESCRIPTION:
Design: multicentric Aims of this study: to describe clinical and genetic basis of Joubert syndrome and cerebello-oculo-renal syndromes.Joubert syndrome (JS) is characterized by hypotonia, abnormal ocular movements and neonatal breathing dysregulation evolving into developmental delay, ataxia, oculomotor apraxia with variable mental retardation. The neuroradiological hallmark of JS is a complex midbrain-hindbrain malformation consisting of vermis hypoplasia/dysplasia, a deepened interpeduncular fossa, and thickened, elongated and mal-orientated superior cerebellar peduncles (Molar Tooth Sign, MTS). Other organs could be involved in JS (kidneys :nephronophthisis or cystic dysplastic kidneys; eyes : Leber Congenital Amaurosis, retinopathy, colobomas); liver : hepatic fibrosis; others: polydactyly, tongue hamartomas, situs inversus). Several associated central nervous system malformations were described : polymicrogyria, hydrocephalus, corpus callosum anomalies and encephalocele. This pleiotropic involvement identifies a large spectrum of cerebello-oculo-renal syndromes or JS Related Disorders (JSRD).

Joubert syndrome and cerebello-oculo-renal syndromes (JS/CORS) are autosomal recessive conditions associated with a high risk of recurrence for further pregnancies (25%). In 2004 mutations in AHI1 gene (Abelson helper integration site gene) were identified in 7-11% JS but the disease is caracterized by a wide genetic heterogeneity. At least five others genes are involved in JS/CORS : NPHP1, which homozygous deletions are responsible for a small percentage of JS (2%) and more recently CEP290 gene which exact mutations prevalence remained to be evaluated.

Using molecular analysis of those three genes (sequencing of 29 coding exons of AHI1 and 54 exons of CEP290, searching for NPHP1 homozygous deletions by PCR analysis) we project to study respective prevalence of mutations of those three genes and described associated phenotypes in 65 JSCORS patients. This work will allowed to described genotype-phenotypes correlation in JSCORS and to progress in the characterization of the underlying pathogenetic mechanisms. It will be the first step before identification of novel disease genes.

ELIGIBILITY:
Inclusion Criteria:

* Child or adult patients without age maximum
* Affected with JS/CORS défined by neurologic disease with at least one of the following symptoms :

  * neonatal hypotonia or developmental delay (before age 3) or mental retardation (QD<70) (after age 3).
  * Ataxia
  * Oculomotor apraxia
* and on MRI :

  * vermis hypoplasia/agenesia defined by insufficient development of cerebellar vermis.
  * And molar tooth defined by thickened, elongated and mal-orientated superior cerebellar peduncles on axial sections.

Exclusion Criteria:

* Chromosomal anomalies identified by caryotype
* Absence of signature of informed consent.
* Absence of affiliation to social security

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children or adult patients affected with JS/CORS
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the prevalence of AHI1 mutations in Joubert syndrome and cerebello-oculo-renal syndromes (JS/CORS) | At the inclusion visit

SECONDARY OUTCOMES:
Assessment of the prevalence of CEP290 mutations and NPHP1 homozygous deletions in JS/CORS ; Caracterization of mutational spectrum of AHI1, NPHP1, CEP290 genes in JS/CORS ; Evaluation of genotype-phenotype correlation in JS/CORS. | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Lydie BURGLEN, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Trousseau, Paris, France